CLINICAL TRIAL: NCT06557369
Title: A Prospective Proof-of-Concept Clinical Investigation to Evaluate Safety and Effectiveness of reSEES in Patients With Intermediate Age-Related Macular Degeneration
Brief Title: A Clinical Trial Evaluating the Safety and Efficacy of a New Light Combination Therapy Addressing Intermediate AMD
Acronym: retinaSEES-PoC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oculox Technologies SA (Industry)
Collaborators: Latis S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oculox Technologies SA
Record Dates: First submitted 2024-05-24; First posted 2024-08-16 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Intermediate AMD
Keywords: phototherapy; subthreshold; laser; Retina; amd; iAMD; photo biomodulation; hyperthermia; mitochondria; choriocapillaris; Para inflammation; cco; RPE; retinal pigment epithelium; chromophore
MeSH Terms: conditions — Glycogen Storage Disease Type II; Hyperthermia; Myopathy, Central Core

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Therapy - Treated Eye (Experimental): Enrolled eye which will receive the light combined treatment.
  Interventions: Device: reSEES
- Intra-patient Control Eye (No Intervention): Contralateral eye used as control to relatively evaluate safety profile and performance

INTERVENTIONS:
Device: reSEES — The treatment consists of combining SMPL and PBM light therapies to exploit the full advantage of their action. The combination will result in an additive or synergetic effect.
  * Treatment sessions are scheduled for three weeks after enrolment (Loading-Phase).
  * Two visits per week are needed.
  * At the first visit of every treatment week, two treatment sessions will follow each other; PBM is applied at least 15' after SMPL (treatment pairs).
  * Only PBM will be administered during the second visit of every treatment week.
  Patients will receive:
  * 1x SMPL treatment at days 0, 7, and 14 (3 in total),
  * 1x PBM treatment at days 0, 3, 7, 10, 14, and 17 (6 in total)
  Nine treatments will be delivered within three weeks. The study will be concluded with three follow-up visits at 18, 24, and 54 weeks.
  Arms: Combination Therapy - Treated Eye

SUMMARY:
The proposed clinical investigation wants primary to validate the safety of the innovative light therapy approach and in second priority provide insight and confirmations on therapeutic effect.

By combining two clinically standard laser-light treatment, both exhibiting a solid-safe profile: the photothermal and the photobiological techniques; the investigational device (reSEES) wants to explore a completely new therapeutic approach by synergically take advantage of the inherent and already observed clinical performances of the two independent techniques.

DETAILED DESCRIPTION:
*Objectives*

1. The primary objective is to evaluate the safety of the reSEES treatment.
2. The secondary objective is to evaluate the effect of the reSEES treatment on the progression of intermediate AMD.

   * Progression of intermediate AMD will be followed for one year,
   * The contralateral eye will be used as a control to compare and observe relative and absolute progression and rate of progression.

*Other objectives*

* Evaluate the evolution of AMD-induced retinal morphological changes.
* Evaluate changes at the choriocapillaris vascular network and analyse/compare eventual transition to nAMD with natural history.
* Evaluate the effect of reSEES on retina functional parameters.
* Investigate the effect of reSEES on patients' perceived vision, mood, and general well-being.
* Evaluate the usability of the proposed laser console.

*Study Details*

30 patients are planned to be included in the study Enrolled patients will receive treatment on the left or the worst eye, and the fellow eye will be used as a control. Enrolled patients must have both eyes eligible for the study (rf. Inclusion Criteria)

*Measurements & Procedures*

The measurements and procedures will be performed within 52 weeks.

* Total number of visits: 10
* Total number of treatments: 9 General health, medical history, and concomitant medication will be assessed and reported.

Ophthalmic examinations will be carried out at different time points: at screening, on Days 3, 10, and 17, and at the follow-up visits at 18, 24, and 52 weeks from T0 Adverse events and occurring changes in concomitant medication will also be collected for evaluation at every time point.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 50 years of age
* Intermediate AMD, Grade AREDS 3
* Both eyes eligible for the study Patients willing to enrol in a clinical study must sign a written informed consent form, cooperate with protocols, and comply with follow-up.
* Dietary supplements and life-style habits must remain unchanged, as far as possible, for the duration of investigation participation.

Exclusion Criteria:

* Myopia > 8D
* Maximum pupillary aperture ᴓ4mm with medical dilation
* Anticipation of ocular surgery during the study
* Clinically significative cataract
* Ocular surgery 6 months or less before study entry
* No previous retinal treatment, neither anti-VEGF (Anti-Vascular Endothelial Growth Factor ) therapy nor laser photocoagulation
* Diabetic retinopathy
* Any other maculopathy and conditions as e.g. retinitis pigmentosa, DME (diabetic macular oedema), retinal lesions, retinal vessel occlusions etc
* Another obfuscating ocular disease including amblyopia, uncontrolled IOP (intraocular pressure), uncontrolled glaucoma or glaucomatous visual field loss, media opacity such as visually significant cataract, epiretinal membrane, vitreomacular traction, etc
* Concomitant systemic diseases and factors affecting the study, as per investigator's discretion
* Pregnant and lactating woman
* Concomitant participation in another interventional clinical study
* When it is expected that the patient will not be able to complete the trial due to mental health, age, or other personal issues.
* Photosensitivity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Absence of autofluorescence (FAF) laser-light spot | From Screening (T0 - 14 days), at each Treatment Sessions (T0, T0 + 3 days, T0 + 7 days, T0 + 10 days, T0 + 14 days, T0 + 17 days), and on all Follow-up Visits (T0 + 18 weeks, T0 + 24 weeks, T0 + 52 weeks)
  Assessment of autofluorescence laser-light spot
Absence of NIR-cSLO laser-light spot traces | From Screening (T0 - 14 days), at each Treatment Sessions (T0, T0 + 3 days, T0 + 7 days, T0 + 10 days, T0 + 14 days, T0 + 17 days), and on all Follow-up Visits (T0 + 18 weeks, T0 + 24 weeks, T0 + 52 weeks)
  Assessment of NIR-cSLO laser-light spot
Treatment-Emergent Adverse Events (TEAE) | From the first Treatment Session (T0), at each subsequent Treatment Sessions (T0 + 3 days, T0 + 7 days, T0 + 10 days, T0 + 14 days, T0 + 17 days), and on all Follow-up Visits (T0 + 18 weeks, T0 + 24 weeks, T0 + 52 weeks)
  Incidence, severity and time of AE

SECONDARY OUTCOMES:
Improvement in visual acuity | From Screening (T0 - 14 days), every second Treatment Sessions (T0 + 3 days, T0 + 10 days, T0 + 17 days), and on all Follow-up Visits (T0 + 18 weeks, T0 + 24 weeks, T0 + 52 weeks)
  Improvement in BCVA
Progression to advanced AMD (SD-OCT) | From Screening (T0 - 14 days), every second Treatment Sessions (T0 + 3 days, T0 + 10 days, T0 + 17 days), and on all Follow-up Visits (T0 + 18 weeks, T0 + 24 weeks, T0 + 52 weeks)
  Rate of progression to advanced AMD by GA area measure
Progression of drusen cross-section (SD-OCT) | From Screening (T0 - 14 days), every second Treatment Sessions (T0 + 3 days, T0 + 10 days, T0 + 17 days), and on all Follow-up Visits (T0 + 18 weeks, T0 + 24 weeks, T0 + 52 weeks)
  Rate of progression of drusen area

OTHER OUTCOMES:
Hyper-Iso-Hypo autofluorescence (FAF - Qualitative Signal Evolution) | From Screening (T0 - 14 days), at each Treatment Sessions (T0, T0 + 3 days, T0 + 7 days, T0 + 10 days, T0 + 14 days, T0 + 17 days), and on all Follow-up Visits (T0 + 18 weeks, T0 + 24 weeks, T0 + 52 weeks)
  Assess the development of the Hyper-Iso-Hypo autofluorescence signal at the perimeter of the GA lesion
Choriocapillaris network reaction (OCTA - Qualitative Signal Evolution) | From Screening (T0 - 14 days), and on all Follow-up Visits (T0 + 18 weeks, T0 + 24 weeks, T0 + 52 weeks)
  Development of the choriocapillaris network
Contrast sensitivity function (Quantitative Pelli-Robson protocol) | From Screening (T0 - 14 days), every second Treatment Sessions (T0 + 3 days, T0 + 10 days, T0 + 17 days), and on all Follow-up Visits (T0 + 18 weeks, T0 + 24 weeks, T0 + 52 weeks)
  Assess visual functions with contrast sensitivity standard tests
Microperimetry | From Screening (T0 - 14 days), and on every second Follow-up Visits (T0 + 18 weeks, T0 + 52 weeks)
  Assessing retinal sensitivity in correspondence of morphological alteration
Perceived vision and mood | From Screening (T0 - 14 days), every second Treatment Sessions (T0 + 3 days, T0 + 10 days, T0 + 17 days), and on all Follow-up Visits (T0 + 18 weeks, T0 + 24 weeks, T0 + 52 weeks)
  Assessment of perceived vision and mood using visual function questionnaire VFQ-25
Usability | At last Treatment Session (T0 + 17 days)
  Assessment of usability of reSEES through questionnaire following standard scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Mario Romano, Prof., Principal Investigator — Director Department of Ophthalmology and Operational Unit, Full professor - Humanitas Gavazzeni
Locations (1):
- Humanitas Castelli, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No